CLINICAL TRIAL: NCT02231489
Title: A Single-Dose, Open Label, Randomized, Two-Way Crossover Pharmacokinetic Study to Assess the Relative Bioavailability of Orally Administered JNJ-42756493 Following Intake of Tablet Versus Capsule in Healthy Subjects
Brief Title: Study to Assess the Relative Bioavailability of Orally Administered JNJ-42756493 Tablet Versus JNJ-42756493 Capsule in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR105269; 42756493EDI1003 (Other: Janssen Research & Development, LLC); 2014-002635-33 (EudraCT Number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42756493; JNJ-61818549
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive treatment A (JNJ-42756493 tablet 10 milligram [mg] as single oral dose) along with JNJ-61818549, 100 microgram (mcg) intravenous infusion over 5 minutes, 2 hours after administration of JNJ-42756493 tablet on Day 1 in Treatment Period 1. Participants will receive treatment B (JNJ-42756493 capsule 10 mg as single oral dose) on Day 1 of Treatment Period 2.
  Interventions: Drug: JNJ-42756493 Tablet; Drug: JNJ-42756493 Capsule; Drug: JNJ-61818549
- Treatment Sequence BA (Experimental): Participants will receive treatment B (JNJ-42756493 capsule 10 mg as single oral dose) along with 100 microgram (mcg) intravenous infusion over 5 minutes, 2 hours after administration of JNJ-42756493 capsule on Day 1 in Treatment Period 1. Participants will receive treatment A (JNJ-42756493 tablet as single oral dose) on Day 1 of Treatment Period 2.
  Interventions: Drug: JNJ-42756493 Tablet; Drug: JNJ-42756493 Capsule; Drug: JNJ-61818549

INTERVENTIONS:
Drug: JNJ-42756493 Tablet — Participants will receive 10 mg of JNJ-42756493 tablet as single oral dose on Day 1 of each treatment period.
Drug: JNJ-42756493 Capsule — Participants will receive 10 mg of JNJ-42756493 capsule as single oral dose on Day 1 of each treatment period.
Drug: JNJ-61818549 — Participants will JNJ-61818549, 100 microgram (mcg) intravenous infusion over 5 minutes, after 2 hours of administration of JNJ-42756493 tablet/capsule on Day 1 Treatment Period 1.

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of JNJ-42756493 oral dose of capsule (reference) versus tablet (test) in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized (study drug assigned by chance), open-label (all people know the identity of the intervention), 2 way crossover (method used to switch participants from one study group change to treatment group), single-dose study in healthy participants. The study will consist of 3 phases: Screening Phase (Day -21 to Day -2), Treatment Phase (consists of 2 single-dose treatment period, either JNJ-42756493 capsule or JNJ-42756493 tablet) and Follow-up Phase (12-14 days after last dose). All the eligible participants will be randomly assigned to 1 of the 2 treatment sequences to ensure that they receive both of the treatments, 1 in each period. Each treatment regimen will be separated by a washout period of at least 15 days. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Relative bioavailability of two dosage form of JNJ-42756493 (test and reference) will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received a thorough explanation of the optional pharmacogenomic research component of the study and was offered an opportunity to participate by signing the separate pharmacogenomic informed consent document
* Female participants must be postmenopausal (no spontaneous menses for at least 2 years, or surgically sterile and must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at screening
* Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator (for example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Participant must have body mass index (BMI) (weight [kilogram {kg}]/height^2 [m^2]) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kg
* Participants must be non-smoker for at least 6 months before entering the study

Exclusion Criteria:

* Participants with a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, metabolic bone disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants with history or current evidence of ophthalmic disorder, such as central serous retinopathy or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Participants with the use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* Participants with positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, hallucinogens or barbiturates at screening and on Day-1 of the first treatment period
* Participants with clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator. Retesting of abnormal lab values that may lead to exclusion will be allowed once

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability (F[abs]) of JNJ-42756493 | Pre-dose;15,30,60,120,130,140,150 and 165 minutes (min),3,4,6,8,12,24,32,48,72,96,120, 144 hours (hrs) post-dose on Day 1 in Treatment Period 1; pre-dose;, 0.25,0.5,1,2,3,4,6,8,12,24,32,48,72,96,120,144 post-dose on Day 1 in Treatment Period 2
  The F (abs) is the percentage of the orally administered dose that is systemically available. It is calculated as (AUC [0-infinity] for test)/(AUC [0-infinity] for reference [ref])*(D for ref/D for test )*100, where the reference treatment is an intravenous administration, AUC (0-infinity) is area under the concentration-time curve from time zero to extrapolated infinite time, and D is the dose of orally administered drug.
Relative Bioavailability (F[rel]) of JNJ-42756493 | Pre-dose;15,30,60,120,130,140,150 and 165 minutes (min),3,4,6,8,12,24,32,48,72,96,120, 144 hours (hrs) post-dose on Day 1 in Treatment Period 1; pre-dose;, 0.25,0.5,1,2,3,4,6,8,12,24,32,48,72,96,120,144 post-dose on Day 1 in Treatment Period 2
  The F (rel) is the percentage of the orally administered dose that is systemically available. It is calculated as (AUC [0-infinity] for test)/(AUC [0-infinity] for reference [ref])*(D for test/D for ref )*100, where the reference treatment is an intravenous administration, AUC (0-infinity) is area under the concentration-time curve from time zero to extrapolated infinite time, and D is the dose of orally administered drug.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-42756493 | Pre-dose;15,30,60,120,130,140,150 and 165 minutes (min),3,4,6,8,12,24,32,48,72,96,120, 144 hours (hrs) post-dose on Day 1 in Treatment Period 1; pre-dose;, 0.25,0.5,1,2,3,4,6,8,12,24,32,48,72,96,120,144 post-dose on Day 1 in Treatment Period 2
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) | Pre-dose;15,30,60,120,130,140,150 and 165 minutes (min),3,4,6,8,12,24,32,48,72,96,120, 144 hours (hrs) post-dose on Day 1 in Treatment Period 1; pre-dose;, 0.25,0.5,1,2,3,4,6,8,12,24,32,48,72,96,120,144 post-dose on Day 1 in Treatment Period 2
  Time to reach the maximum plasma JNJ4-2756493 concentration.
Elimination Half-Life (t [1/2] Lambda) | Pre-dose;15,30,60,120,130,140,150 and 165 minutes (min),3,4,6,8,12,24,32,48,72,96,120, 144 hours (hrs) post-dose on Day 1 in Treatment Period 1; pre-dose;, 0.25,0.5,1,2,3,4,6,8,12,24,32,48,72,96,120,144 post-dose on Day 1 in Treatment Period 2
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium